CLINICAL TRIAL: NCT02033083
Title: Laminaria Compared to Dilapan-S for Cervical Preparation Before Dilation and Evacuation at 18-24 Weeks of Gestation: A Randomized Controlled Trial
Brief Title: Laminaria Compared to Dilapan-S for Cervical Preparation Before Dilation and Evacuation at 18-24 Weeks of Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of Greater New York (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: laminariavsdilapan
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Second Trimester Abortion
Keywords: abortion; cervical dilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laminaria (Active Comparator): Patients in this arm will receive laminaria cervical dilators one day before D&E procedure.
  Interventions: Device: Laminaria
- Dilapan-S (Active Comparator): Patients in this arm will receive Dilapan-S cervical dilators one day before D&E procedure.
  Interventions: Device: Dilapan-S

INTERVENTIONS:
Device: Laminaria
  Arms: Laminaria
Device: Dilapan-S
  Arms: Dilapan-S

SUMMARY:
Primary objective: To study the difference in dilation and evacuation (D&E) procedure time following overnight cervical preparation with laminaria or Dilapan-S™. The investigators hypothesize procedure time will be less with Dilapan-S™.

Secondary objectives: To compare the use of laminaria and Dilapan-S™ for differences in: (1) initial cervical dilation before D&E; (2) need for mechanical dilation to accomplish D&E and ease of dilation if required; (3) number of osmotic dilators placed; (4) ability to complete the D&E procedure without further cervical preparation; (5) complications; (6) pain and other side effects; (7) patient acceptability; and (8) provider acceptability.

DETAILED DESCRIPTION:
One hundred eighty women were randomized evenly across treatment arms, stratified by gestational age groups of 18 0/7-20 6/7 (n= 91) and 21 0/7-24 0/7 (n=87). The analytic sample N=173 (laminaria=86, Dilapan=87); 2 cases were removed for post-randomization exclusion and 5 for missing data on one or more outcome variables. Demographic information and results for the primary outcome of procedure time are reported below in tabular form in the results section.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Seeking pregnancy termination from 18 0/7 to 24 0/7 weeks of gestation
* Eligible for pregnancy termination at Planned Parenthood of New York City
* Able to give informed consent
* English speaking

Exclusion Criteria:

* • Active bleeding or hemodynamically unstable at enrollment

  * Signs of chorioamnionitis or clinical infection at enrollment
  * Signs of spontaneous labor or cervical insufficiency at enrollment
  * Spontaneous intrauterine fetal demise
  * Allergy to laminaria or Dilapan-S™

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Planned Parenthood of New York City
Locations (1):
- Planned Parenthood of New York City, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients identified during surgical abortion services by tracking gestational age using electronic health record. Patients seeking abortion services undergo standard clinical procedures for pre-operative evaluation, and routine abortion counselling and surgical consent. After clinic staff confirmed patient is eligibility, research staff tell her about the study and, if the patient is interested in study participation, screen her for inclusion and exclusion criteria.
Pre-assignment Details: If eligible for study participation, the member of the research team will review study procedures and the risks and benefits of participation with the patient, and obtain informed consent for study participation. Once informed consent is obtained, participants will be assigned a screening number. Research staff will then administer a verbal 10-minute survey (Form 1) to collect demographic information and assess baseline pain, bleeding, nausea and other pregnancy-related symptoms.
Groups:
- Laminaria: Patients in this arm will receive laminaria cervical dilators one day before D&E procedure.
  Laminaria
- Dilapan-S: Patients in this arm will receive Dilapan-S cervical dilators one day before D&E procedure.
  Dilapan-S
Period: Overall Study
Arm/Group | Laminaria | Dilapan-S
Started | 90 | 90
Completed | 89 | 89
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laminaria | Dilapan-S | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.99 (4.49) | 23.80 (4.61) | 23.90 (4.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 89 | 178
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American or Black | 42 | 45 | 87
  Hispanic or Latina | 21 | 18 | 39
  White | 8 | 16 | 24
  Other | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: D&E Procedure Time
Description: Length of D&E procedure in minutes
Time Frame: The primary outcome measure will be assessed on the day of the patient's D&E procedure. (day 2)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Laminaria | Dilapan-S
Number analyzed (Participants) | 88 | 88
minutes | 7.35 (3.63) | 7.55 (4.59)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Laminaria | Dilapan-S
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 0/89 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No